CLINICAL TRIAL: NCT02728895
Title: An Open-Label, Dose-Finding Study of Vedolizumab IV Plus Standard of Care for Graft-Versus-Host Disease (GvHD) Prophylaxis in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Dose Finding Study of Vedolizumab for GvHD in Participants Undergoing Allogeneic HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-1015; U1111-1184-1822 (Registry Identifier: WHO)
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-07

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation
Keywords: Drug Therapy
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Vedolizumab 75 mg (Experimental): Vedolizumab 75 mg, injection, intravenously once on Days -1, 13 and 42.
  Interventions: Drug: Vedolizumab
- Cohort 2: Vedolizumab 300 mg (Experimental): Vedolizumab 300 mg, injection, intravenously once on Days -1, 13 and 42.
  Interventions: Drug: Vedolizumab
- Cohort 3: Vedolizumab Dose 1 (Experimental): Vedolizumab first decided dose as determined from Cohort 1 or 2, injection, intravenously once on Days -1, 13 and 42.
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab Injection.

SUMMARY:
The purpose of this study is to assess the initial tolerability, safety and recommended phase 2 dose of vedolizumab intravenous (IV) administered for GvHD prophylaxis along with standard GvHD prophylaxis therapy (in participants undergoing allogeneic hematopoietic stem cell transplantation [allo-HSCT]).

DETAILED DESCRIPTION:
The drug being tested in this study is called Vedolizumab. Vedolizumab (also called MLN0002) is approved for the treatment of adult participants with moderately to severely active ulcerative colitis (UC) and Crohn's disease (CD) who achieved an inadequate response, had a loss of response, or were intolerant to conventional and/or biologic treatments. This study will look at the tolerability and pharmacokinetics of Vedolizumab in participants undergoing allo-HSCT when added to standard GvHD prophylaxis (tacrolimus plus short-term methotrexate) for the prevention of acute GvHD (major complication in allo-HSCT).

The study will enroll approximately 36 participants. Participants will be assigned to different dose-escalating cohorts in order to find out the recommended phase 2 dose (RP2D) of the study:

* Cohort 1: Vedolizumab 75 mg
* Cohort 2: Vedolizumab 300 mg
* Cohort 3: Vedolizumab Dose 1

All participants have to receive 1 injection of Vedolizumab on Day -1 before allo-HSCT and on Days 13 and 42 after allo-HSCT. If none of the participants receiving vedolizumab at 75 mg experience dose-limiting toxicities (DLTs), dose escalation will continue to 300 mg on Day -1 before allo-HSCT and on Days +13 and +42 after allo-HSCT. If the first 3 participants at 300 mg tolerate the treatment without experiencing DLTs, then the decision on whether to increase the vedolizumab IV dose in the next cohort will be guided by the PK results.

Cohorts will be escalated in same manner until the identification of RP2D. The cohort at that dose level may be expanded to include approximately 18 additional participants undergoing myeloablative conditioning or reduced-intensity conditioning (RIC) and receiving either related or unrelated allo-HSCT for the treatment of hematologic malignancies or myeloproliferative neoplasms. This group of participants will allow the further assessment of the tolerability and clinical activity of vedolizumab.

This multi-center trial will be conducted in the United States. The overall time to participate in this study will be approximately 2 years. Following the treatment period, participants who remain in remission will be followed for development of acute and chronic GvHD and safety during clinic visits at 4, 5, 6, 9, and 12 months after allo-HSCT or until death or withdrawal of consent or termination of the study by the sponsor. Participants who complete the study will attend a 12-month follow-up visit. Patients who have been discontinued from treatment will attend an end of treatment visit 30 to 40 days after the last dose of study drug using all study procedures outlined for the 12-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Is undergoing matched or single-antigen mismatched unrelated-donor myeloablative transplant for the treatment of acute lymphoblastic leukemia (ALL) or acute myeloid leukemia (AML); Is less than or equal to (<=) 60 years of age.

   For the cohort after RP2D
2. Is undergoing matched or single-antigen mismatched related or unrelated-donor transplant and receiving myeloablative conditioning or RIC for the treatment of hematologic malignancies or myeloproliferative neoplasms; Is less than or equal to (<=) 75 years of age.

Exclusion Criteria:

1. Has received prior allogeneic transplants or who are planned to undergo umbilical cord blood transplant, receive ex vivo T-cell-depleted hematopoietic stem cells (HSCs), received any in vivo T-cell depleting antibodies, or non-myeloablative conditioning.
2. Has active cerebral/meningeal disease, active cytomegalovirus (CMV) colitis, or signs and symptoms of progressive multifocal leukoencephalopathy (PML) or any history of PML.
3. Is undergoing transplant for the treatment of nonmalignant hematological disorders (for example: aplastic anemia, sickle cell anemia, thalassemias, Fanconi anemia).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - OSU - James Comprehensive Cancer Center, Columbus, Ohio
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Chen YB, Shah NN, Renteria AS, Cutler C, Jansson J, Akbari M, Chen C, Quadri S, Parfionovas A, Devine SM. Vedolizumab for prevention of graft-versus-host disease after allogeneic hematopoietic stem cell transplantation. Blood Adv. 2019 Dec 10;3(23):4136-4146. doi: 10.1182/bloodadvances.2019000893. PMID 31821456

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 15 June 2016 to 10 July 2018.
Pre-assignment Details: Participants undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT) were enrolled to receive vedolizumab intravenous 75 milligram (mg) or 300 mg along with standard graft-versus-host disease (GvHD) prophylaxis therapy (tacrolimus plus short team methotrexate).
Groups:
- Cohort 1: Vedolizumab 75 mg: Vedolizumab 75 mg, 30-minutes infusion, intravenously, once on Day -1 (before allo-HSCT on Day 1), and Days 13 and 42 (after allo-HSCT on Day 1).
- Cohort 2: Vedolizumab 300 mg: Vedolizumab 300 mg, 30-minutes infusion, intravenously once on Days -1 (before allo-HSCT on Day 1), and Days 13 and 42 (after allo-HSCT on Day 1).
Period: Overall Study
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Started | 3 | 21
Completed | 2 | 16
Not Completed | 1 | 5
Not completed — Other | 1 | 2
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Population: The population of participants evaluable for vedolizumab safety was defined as all participants who received any amount of vedolizumab intravenously.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg | Total
Number analyzed (Participants) | 3 | 21 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (17.44) | 52.7 (16.90) | 49.9 (18.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 1 | 16 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 18 | 21
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 19 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 21 | 24
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 92.93 (25.662) | 89.96 (25.836) | 90.33 (25.272)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLTs was based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and was defined as any of following events: Grade 3 or higher toxicity assessed by the investigator as related to vedolizumab treatment; Grade 4 or higher regimen-related organ toxicities; and failure to engraft by Day +28. Engraftment was defined as absolute neutrophils count (ANC) greater than (>) 500 per cubic millimeter (/mm^3) for 3 consecutive days or >2000/mm^3 for 1 day.
Time Frame: Baseline up to Day 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
Participants | 0 | 0

2. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to 18 weeks after last dose of study drug
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
Participants
  TEAEs | 3 | 21
  SAEs | 2 | 11

3. Primary Outcome: Mean Serum Concentrations of Vedolizumab That Helped the Likelihood of Alpha4Beta7 Target Saturation on Day 100 Following Allo-HSCT
Time Frame: Day 100
Population: The pharmacokinetic (PK) population was defined as participants from the safety set with at least 1 PK sample collected. The PK population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 2 | 18
microgram per milliliter (mcg/mL) | 7.34 (3.762) | 18.36 (11.043)

4. Secondary Outcome: Time to Neutrophil Engraftment
Description: Time to neutrophil engraftment (recovery of ANC) was defined by an ANC >500/mm^3 for 3 consecutive days or >2000/mm^3 for 1 day. Time to neutrophil engraftment was calculated using Kaplan-Meier estimate and presented with 2-sided 95% confidence interval.
Time Frame: Baseline up to Day 100
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
days | 22 [15 to 22] | 14 [13 to 17]

5. Secondary Outcome: Percentage of Participants With Overall Grade 2 to 4 Acute Graft-Versus-Host Disease (GvHD)
Description: GvHD grading scale was based on the modified Glucksberg criteria. The grades are defined as: Grade 1 (skin stage 1 or 2 only); Grade 2 (skin stage 3 or liver stage 1 or lower or gastrointestinal [GI] stage 1 or upper GI involvement); Grade 3 (skin stage 0 to 3 plus liver stage 2 to 4 or lower GI stage 2 to 3); Grade 4 (skin stage 4 or lower GI stage 4).
Time Frame: Baseline up to Day 100
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
percentage of participants | 0 [0 to 70.8] | 19.0 [5.4 to 41.9]

6. Secondary Outcome: Percentage of Participants With Maximum Severity of Acute GvHD Based on Modified Glucksberg Criteria
Description: Maximum severity was assessed using GvHD grading scale based on the modified Glucksberg criteria. The grades are defined as: Grade 1 (skin stage 1 or 2 only); Grade 2 (skin stage 3 or liver stage 1 or lower or GI stage 1 or upper GI involvement); Grade 3 (skin stage 0 to 3 plus liver stage 2 to 4 or lower GI stage 2 to 3); Grade 4 (skin stage 4 or lower GI stage 4).
Time Frame: Baseline up to Day 100
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
percentage of participants
  Grade 1 | 66.7 [17.5 to 95.0] | 28.6 [11.3 to 55.6]
  Grade 2 | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade 2 severity. | 14.3 [3.8 to 41.1]
  Grade 3 | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade 3 severity. | 4.8 [0.6 to 29.7]
  Grade 4 | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade 4 severity. | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade 4 severity.

7. Secondary Outcome: Percentage of Participants With Maximum Severity of Acute GvHD Based on Blood and Marrow Transplant Clinical Trials Network (BMT CTN) Modified International Bone Marrow Transplant Registry Database (IBMTR) Index
Description: Maximum severity of acute GvHD was assessed by using BMT CTN modified IBMTR index. The severity index are defined as: Grade A (skin stage 1: extent of rash less than [<] 25%); Grade B (skin stage 2: extent of rash 25 to 50% or liver stage 1 to 2: total bilirubin 34 to 102 micromole per liter [mcmol/L] or intestinal tract stage 1 to 2: volume of diarrhea 550 to 1500 milliliter per day [mL/day]); Grade C (skin stage 3: extent of rash greater than (>) 50% or liver stage 3: total bilirubin 103 to 255 mcmol/L or intestinal tract stage 3: volume of diarrhea >1500 mL/day); Grade D (skin stage 4: extent of rash bullae or liver stage 4: total bilirubin >255 or intestinal tract stage 4: volume of diarrhea severe pain and ileus).
Time Frame: Baseline up to Day 100
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
percentage of participants
  Grade A | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade A severity. | 19.0 [6.1 to 46.2]
  Grade B | 66.7 [17.5 to 95.0] | 14.3 [3.8 to 41.1]
  Grade C | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade C severity. | 14.3 [3.8 to 41.1]
  Grade D | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade D severity. | 0 [NA to NA] — Upper limit and lower limit of confidence interval could not be calculated because no participants had Grade D severity.

8. Secondary Outcome: Ctrough: Serum Concentration Before Dosing for Vedolizumab
Time Frame: Days 13 and 42 pre-dose
Population: The PK population was defined as participants from the safety set with at least 1 PK sample collected. The PK population where data at specified time points was available.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
Number analyzed (Participants) | 3 | 21
mcg/mL
  Day 13 | 5.87 (3.00) | 21.34 (6.05)
  Day 42: number analyzed (Participants) | 3 | 19
  Day 42 | 8.17 (5.20) | 29.05 (13.04)

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug and no more than Week 18 after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1: Vedolizumab 75 mg | Cohort 2: Vedolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/21
Serious Adverse Events (participants affected / at risk) | 2/3 | 11/21
Other Adverse Events (participants affected / at risk) | 3/3 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Vedolizumab 75 mg (N=3) | Cohort 2: Vedolizumab 300 mg (N=21)
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Embolism (Vascular disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Vedolizumab 75 mg (N=3) | Cohort 2: Vedolizumab 300 mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 1 | 5
Sinus bradycardia (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 13
Nausea (Gastrointestinal disorders) | 1 | 12
Stomatitis (Gastrointestinal disorders) | 3 | 10
Vomiting (Gastrointestinal disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anorectal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 3 | 12
Pyrexia (General disorders) | 2 | 11
Oedema peripheral (General disorders) | 0 | 5
Oedema (General disorders) | 0 | 4
Chills (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 1
Chronic graft versus host disease (Immune system disorders) | 0 | 1
Chronic graft versus host disease in skin (Immune system disorders) | 0 | 1
Engraftment syndrome (Immune system disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 4
Clostridium difficile infection (Infections and infestations) | 0 | 3
Candida infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin candida (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 1
Vulvitis (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 2 | 15
Neutrophil count decreased (Investigations) | 1 | 10
White blood cell count decreased (Investigations) | 2 | 7
Alanine aminotransferase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 6
Blood creatinine increased (Investigations) | 1 | 6
Lymphocyte count decreased (Investigations) | 1 | 6
Blood bilirubin increased (Investigations) | 1 | 4
Haemoglobin decreased (Investigations) | 1 | 3
Weight decreased (Investigations) | 0 | 4
Hepatic enzyme increased (Investigations) | 0 | 2
Bacterial test positive (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Clostridium test positive (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Enterococcus test positive (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 17
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 9
Dysgeusia (Nervous system disorders) | 1 | 4
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Tremor (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 3
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Product contamination microbial (Product Issues) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 1 | 1
Agitation (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 2
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Scrotal erythema (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 6
Hypotension (Vascular disorders) | 0 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT02728895/SAP_000.pdf
  • Study Protocol (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT02728895/Prot_001.pdf